CLINICAL TRIAL: NCT06786533
Title: Phase 1 Study of Anti-FLT3 Chimeric Antigen Receptor-redirected T Cells in Subjects With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Clinical Study of Anti-FLT3 CAR-T Cells for the Treatment of Relapsed/Refractory AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hemogenyx Pharmaceuticals LLC (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HEM-001-AML-1101; IND 029573 (Other: FDA)
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose and route of administration HG-CT-1 cells will be administered by intravenous infusion following standard lymphodepleting chemotherapy consisting of fludarabine and cyclophosphamide.
  Statistical Design The trial will use a modified toxicity probability interval (mTPI-2) design while matching the cohort size with the traditional 3 + 3 design.
  Dose Levels Dose level 1: 7x10^7 Transduced CAR+ HG-CT-1 Dose level 2: 1.4x10^8 Transduced CAR+ HG-CT-1 Dose level 3: 3.5x10^8 Transduced CAR+ HG-CT-1 If Dose level 1 is found not to be safe, dose will be de-escalated to 3.5 x 10^7 Transduced CAR+ HG-CT-1. (Dose level -1)
  Pediatric Dosing:
  Enrollment on any pediatric (≥12 and <18 years of age) cohort shall begin after the corresponding adult cohort has been safely completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose level 1: 7x10^7 Transduced CAR+ HG-CT-1 (Experimental)
  Interventions: Drug: Anti-FLT3 CAR-T cells
- Dose level 2: 1.4x10^8 Transduced CAR+ HG-CT-1 (Experimental)
- Dose level 3: 3.5x10^8 Transduced CAR+ HG-CT-1 (Experimental)
  Interventions: Drug: Anti-FLT3 CAR-T cells
- Dose level -1: 3.5 x 10^7 Transduced CAR+ HG-CT-1 (Experimental)
  Interventions: Drug: Anti-FLT3 CAR-T cells

INTERVENTIONS:
Drug: Anti-FLT3 CAR-T cells — Anti-FLT3 CAR-T cells is administered by intravenous infusion following standard lymphodepleting chemotherapy consisting of fludarabine and cyclophosphamide.
  Other Names: HG-CT-1
  Arms: Dose level -1: 3.5 x 10^7 Transduced CAR+ HG-CT-1; Dose level 1: 7x10^7 Transduced CAR+ HG-CT-1; Dose level 3: 3.5x10^8 Transduced CAR+ HG-CT-1

SUMMARY:
This is a phase 1 dose escalation study to determine the safety of anti-FLT3 CAR-T in subjects with R/R AML. The primary objective is to assess safety. Up to 18 evaluable adult and 18 evaluable pediatric subjects will be enrolled. Evaluable subjects are defined as those who have received an infusion of HG-CT-1.

Primary clinical objectives:

i. Determine the safety of HG-CT-1 based on the proportion of subjects infused with HG-CT-1 who experience a dose limiting toxicity (DLT).

Secondary clinical objectives:

i. Estimate the efficacy of HG-CT-1 according to standard clinical response criteria for AML.

ii. Estimate overall survival of evaluable subjects. iii. Estimate progression-free survival of evaluable subjects. iv. Estimate duration of response in evaluable subjects who achieve a response.

Secondary scientific objectives:

i. Describe the persistence and trafficking of HG-CT-1. ii. Describe HG-CT-1 bioactivity and its predictors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at enrollment. Patients ≥12 and <18 12 to 17 years of age weighing ≥ 35 kg at enrollment may be included once safety evaluation at the corresponding adult dose escalation protocol have been completed.
* Subjects with AML unlikely to be cured with currently available therapies. Specifically, the following groups are eligible:

  1. Refractory AML: i.e., newly diagnosed AML that after two cycles of intensive chemotherapy has not achieved a complete remission or morphologic leukemia free state by ELN criteria.1 Intensive chemotherapy must have included either the combination of cytarabine and an anthracycline (7+3 or similar) or combination of venetoclax with a hypomethylating agent.

     Patients with FLT3 ITD must also have failed treatment with a FLT3 inhibitor and patients with IDH1 or IDH2 mutations must have failed treatment containing ivosidenib or enasidenib respectively (i.e., progression on treatment, or failure to achieve CR after six months of treatment,) OR:
  2. AML relapsed following allogeneic stem cell transplantation (including MDS evolved to AML post-allogeneic stem cell transplantation). Note: morphologic relapse is not required; persistent/recurrent disease-associated molecular, phenotypic, or cytogenetic abnormalities (measurable residual disease, MRD) at any time after allogeneic HSCT is eligible. OR:
  3. AML that has relapsed within 12 months after initial induction and consolidation therapy OR:
  4. AML that has relapsed more than 12 months after initial induction but that has failed to achieve CR or morphologic leukemia free state after one reinduction OR:
  5. AML after second or subsequent relapse.
* FLT3 expression must be detectable in AML blast by flow cytometric analysis.
* Subjects must have a suitable stem cell transplant donor. Donor may be matched or mismatched and must be found to be suitable according to the institution's standard criteria. That donor shall be "cleared" for donation by institutional standards prior to administration of HG-CT-1. Adult donors can be either related or unrelated, HLA-matched or partially matched. Matched or partially matched umbilical cord blood donors are also eligible.
* Subjects with relapsed disease after prior allogeneic transplant must be off systemic immunosuppression for at least 1 month at the time of enrollment without GvHD that requires systemic immunosuppression.
* Satisfactory organ functions:

  1. Creatinine ≤ 1.6 mg/dl and Creatinine clearance (CrCl) as calculated by the Cockcroft-Gault formula ≥ 60 mL/min.
  2. ALT/AST must be ≤ 3 x upper limit of normal unless related to disease.
  3. Direct bilirubin < 2.0mg/dl unless subject has Gilbert's syndrome (in which case it should be ≤3.0 mg/dL).
  4. Left ventricular ejection fraction ≥ 45% as confirmed by echocardiogram or MUGA.
  5. DLCO >45% predicted and O2 Saturation > 90% on room air.
* Patients ≥18 must have an ECOG Performance status 0-1. Patients <18 must have a Lansky/Karnofsky score of ≥50.
* Written informed consent is given in patients ≥ 18. In patients <18 or not developmentally appropriate for consent, written consent will be provided to the parent or legal guardian. Patients ≥12 and <18 years of age will be additionally provided with assent documentation.
* Subjects of reproductive potential must agree to use acceptable birth control methods (as described in protocol Section 4.7).

Exclusion Criteria:

* Pregnant or lactating (nursing) women.
* Active second malignancy will not be eligible with the following exceptions:

  1. Carcinoma in situ of the cervix (which may be considered for enrollment),
  2. Indolent, non-metastatic prostate cancer
  3. Non melanoma skin cancer
  4. Other indolent and controlled malignancies not requiring urgent treatment.
* Subjects with a history of a prior allogeneic stem cell transplantation are excluded if:

  1. Subjects are less than 100 days post-transplant OR
  2. Subjects have evidence of ongoing active GvHD and are taking immunosuppressive agents (>0.5mg/kg/methylprednisolone equivalents or other immunosuppression for GvHD treatment) OR
  3. Subjects have received DLI within 30 days prior to enrollment.
* Active hepatitis B (HBV) or active hepatitis C (HCV) or any HIV infection. Note: prior HCV that has been appropriately treated or evidence of past HBV infection do not constitute exclusions.
* Concurrent use of systemic steroids at a prednisone dose of greater than 10 mg, hydrocortisone greater than 10-12.5 mg/m2/day, or equivalent. Recent, or current use of inhaled steroids is not exclusionary.
* Concurrent use of immunosuppressant medications such as calcineurin inhibitors, methotrexate, or alemtuzumab.
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the site Pl would pose an unacceptable risk to the subject.
* Active or uncontrolled viral, bacterial, or fungal infection. May be receiving ongoing therapy for controlled infection.
* Subjects with signs or symptoms indicative of active CNS involvement. A CNS evaluation shall be performed as clinically appropriate to rule out CNS involvement. Subjects with adequately treated CNS leukemia are eligible. History of CNS involvement is not exclusionary if CNS has been cleared with a documented negative lumbar puncture and negative imaging (imaging required only if previously showing evidence of CNS leukemia not otherwise documented by spinal fluid assessment).
* Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
* Hyperleukocytosis (>50,000 blasts/µL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy.
* Patients with Acute Promyelocytic Leukemia are not eligible.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of HG-CT-1 cells based on the proportion of subjects infused with HG-CT-1 who experience a DLT. | From the time of HG-CT-1 infusion until Day 28
  Occurrence of dose-limiting toxicities related to HG-CT-1. First-in-human study with unknown safety of infusion of HG-CT-1.

SECONDARY OUTCOMES:
Estimate the efficacy of HG-CT-1 cells as defined by clinical response according to established criteria for AML. | Day 14, Day 28, Month 3, Month 6 and Month 12
  Proportion of subjects with response, according to ELN 2022 criteria. {Dohner et al., 2022 #29518}. To demonstrate the anti-AML activity of HG-CT-1.
Estimate the Overall Survival (OS). | At 6 months and 1 year
  Proportion of subjects alive at 6 months and one year. To demonstrate effect on disease biology and prognosis (compared to historical expectations).
Estimate the progression-free survival (PFS). | At 6 months and 1 year
  Proportion of subjects alive without progression at 6 months and one year. To demonstrate durability of anti-AML effect.
Estimate the Duration of response (DOR). | At 6 months and 1 year
  Proportion of subjects with response who remain alive and without progression at 6 months and at one year. To demonstrate durability of anti-AML effect.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided